CLINICAL TRIAL: NCT02689219
Title: A Multicenter Phase II Study of Brentuximab Vedotin in Relapsed/Refractory Germ Cell Tumors
Brief Title: Brentuximab Vedotin in Relapsed/Refractory Germ Cell Tumors
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding/ benefit
Sponsor: Nabil Adra (Other)
Responsible Party: Sponsor-Investigator, Nabil Adra, Assistant Professor of Clinical Medicine, Indiana University School of Medicine
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IUSCC-0568
Record Dates: First submitted 2016-02-12; First posted 2016-02-23 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Germ Cell Tumors; Testis Cancer; Testicular Cancer; Embryonal Carcinoma; Nonseminomatous Germ Cell Tumor
Keywords: Antigens, CD30, Embryonal Germ Cell Tumors
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Testicular Neoplasms; Carcinoma, Embryonal; Nonseminomatous germ cell tumor | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CD30 positive (Experimental): Brentuximab vedotin, 1.8 mg/kg (1.2 mg/kg in patients with grade 2 peripheral neuropathy at enrollment) will be administered by IV infusion given over approximately 30 minutes on Day 1 of each 21-day cycle.
  Interventions: Drug: Brentuximab Vedotin
- CD30 negative/unknown (Experimental): Brentuximab vedotin, 1.8 mg/kg (1.2 mg/kg in patients with grade 2 peripheral neuropathy at enrollment) will be administered by IV infusion given over approximately 30 minutes on Day 1 of each 21-day cycle.
  Interventions: Drug: Brentuximab Vedotin

INTERVENTIONS:
Drug: Brentuximab Vedotin — Both cohorts will be treated similarly and in parallel but analyzed separately.
  Other Names: SGN-35

SUMMARY:
This is a Phase II study to evaluate the activity of brentuximab vedotin in relapsed/refractory non-seminomatous germ cell tumors (NSGCT).

DETAILED DESCRIPTION:
Primary Objective To determine the anti-tumor efficacy of brentuximab vedotin in relapsed/ refractory NSGCT.

Secondary Objectives

1. To determine the progression free survival in patients with relapsed/ refractory NSGCT treated with brentuximab vedotin.
2. To determine the overall survival of patients with relapsed/ refractory NSGCT treated with brentuximab vedotin.
3. To determine the safety and tolerability of brentuximab vedotin in this patient population.

Eligible patients will be divided into two cohorts, those who are CD30 positive and those who are CD30 negative/unknown. Both groups will be treated similarly and in parallel but analyzed separately. CD30 status may be unknown in the unlikely case of tumor-marker-only relapse or when a fresh tumor biopsy is not feasible, and archival tumor tissue is not obtainable despite efforts to do so. These patients will be included in the CD30 negative cohort for analysis purposes, since statistically NSGCT are more likely to be CD30 negative. The number of such patients with unknown CD30 status should not exceed 5 patients.

Eligible patients will be treated with brentuximab vedotin at 1.8 mg/kg IV every 3 weeks (maximum dose of 180 mg) indefinitely until disease progression, unacceptable toxicity, or study closure.Eligible patients with grade 2 peripheral neuropathy at enrollment will be treated with brentuximab vedotin at 1.2 mg/kg IV every 3 weeks (maximum dose of 180 mg) indefinitely until disease progression, unacceptable toxicity, or study closure. Response to treatment will be assessed clinically with history, physical exam and tumor markers measurement (BHCG and AFP) on day 1 of each cycle and with CT scans after cycle 2, 4, and every 4 cycles thereafter while receiving treatment.

ELIGIBILITY:
Inclusion Criteria

Subject must meet all of the following applicable inclusion criteria to participate in this study:

1. Age ≥ 18 years at the time of informed consent.
2. Patients with histologically or serologically confirmed relapsed/refractory non-seminoma germ cell tumor, (i.e., embryonal carcinoma, choriocarcinoma, or yolk sac tumors) including female GCT and primary mediastinal NSGCT.
3. Patients must have progressed after prior high dose chemotherapy (HDCT) treatment, been deemed not to be a candidate for high dose chemotherapy or refused high-dose chemotherapy, and be considered incurable by other standard therapies including further chemotherapy or surgery. There is no maximum allowable number of previous therapies.

   "Failure" of prior therapy is defined as:
   1. A >25% increase in the products of perpendicular diameters of measurable tumor masses during prior therapy which are not amenable to surgical resection.
   2. The presence of new tumors which are not amenable to surgical resection.
   3. An increase in AFP or beta-hCG (two separate determinations at least one week apart are required if rising tumor markers are the only evidence of failure).

   NOTE: Patients with clinically growing "teratoma" (normal declining tumor markers and radiographic or clinical progression) should be considered for surgery.
4. Patients must have evidence of recurrent or metastatic carcinoma by one or more of the following:

   i) The appearance of metastatic disease by standard imaging techniques ii) The appearance of rising serum tumor marker, AFP or beta-hCG NOTE: If a rising tumor marker is the only evidence of progressive disease, at least 2 consecutive rising values at least one week apart are needed. Patients with only evidence of disease is rising tumor marker AFP and beta-hCG will be provided alternate causes of increased serum levels of these markers are not present, such as cross reaction with luteinizing Hormone (LH) (that can be tested if needed by testosterone suppression of LH), hepatitis, use of marijuana or second primary tumor, etc.
5. Patients with primary medistinal non seminomatous germ cell tumor are eligible if they have received first line platinum based chemotherapy and their recurrence is not amenable to surgical resection based on the treating physician expert opinion.
6. Patients with late relapse (>2 years) of non seminomatous germ cell tumors are eligible if they have received first line platinum based chemotherapy and their recurrence is not amenable to surgical resection based on the treating physician expert opinion.
7. Patients with brain metastases are allowed onto the study as long as patients have completed their treatment for brain metastasis, no longer require corticosteroids, and are asymptomatic. Subjects with neurological symptoms should undergo a head CT scan or brain MRI to exclude brain metastasis, at the discretion of the treating physician.
8. Patients with ECOG performance status of 0-2.
9. Adequate organ and marrow function as defined below:

   1. Hemoglobin ≥ 8 g/dL
   2. Absolute neutrophil count ≥ 1,000/mm3
   3. Platelet count ≥ 75,000/mm3
   4. Total bilirubin ≤ 1.5 × ULN except patients with documented Gilbert's syndrome (≤ 3 × ULN)
   5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN; for patients with hepatic metastases, ALT and AST ≤ 5 × ULN
   6. Calculated creatinine clearance ≥ 30 mL/min as determined by the Cockcroft-Gault equation.
10. Patients who are willing and able to comply with the protocol and study procedures including willingness to undergo tumor biopsy for tumor cells before therapy to assess for CD30 status (unless archival tumor tissue from orchiectomy or other previous sample is not obtainable despite efforts to do so and a fresh tumor biopsy is not feasible).
11. Females of childbearing potential must not be pregnant or breast-feeding. Male and female patients of reproductive potential must agree to use two forms of highly effective contraception from the screening visit through 28 days after the last dose of study drug. Acceptable forms of effective contraception include:

    * Oral, injected or implanted hormonal methods of contraception.
    * Placement of an intrauterine device (IUD) or intrauterine system (IUS).
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
    * Male sterilization (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
    * True abstinence: When this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.] Pregnancy tests for females of childbearing potential are required; must be serum at screening and the post treatment safety assessment visit. A positive urine pregnancy test must be confirmed by a serum pregnancy test and a pelvic US since some NSGCT may secrete beta-hCG and cause a false positive pregnancy. A pelvic US does not need to be repeated with each cycle unless the treating physician thinks it is necessary to do so.
12. Potential subject must have the ability to understand (as judged by the treating physician) and willingness to provide written informed consent and HIPAA authorization for release of personal health information.

NOTE: HIPAA authorization may be included in the informed consent or obtained separately. Written informed consent must be obtained from a potential subject prior to the conduct of any study-specific procedures.

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the study:

1. Patients with pure seminoma.
2. Patients with pure teratoma.
3. Chemotherapy within 2 weeks of initiating study treatment. There is no maximum allowable number of previous therapies.
4. Major surgery within 3 weeks of starting study treatment. There is no minimum time requirement for minor procedures such as biopsy or vascular access placement.
5. Radiation within 2 weeks of starting study treatment.
6. ≥ Grade 3 neuropathy at the time of enrollment.
7. Pregnancy or breast-feeding.
8. Previous treatment with any anti-CD30 directed therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2018-11-13 (Actual); Study Completion 2019-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Costantine Albany, MD, Principal Investigator — Indiana University School of Medicine, Indiana University Simon Cancer Center
Locations (4):
- United States (4):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Memorial Sloan Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was a two cohort Phase II study. A Simon two-stage design was used. One cohort (CD30 negative/unknown) met the stopping rule for lack of efficacy at the first stage interim analysis. The first stage of the second cohort (CD30 positive) was not completed because the study was stopped early due to lack of funding.
Groups:
- CD30 Negative/Unknown: Brentuximab Vedotin 1.8 mg/kg (1.2 mg/kg in patients with grade 2 peripheral neuropathy at enrollment) administered by IV infusion given over approximately 30 minutes on Day 1 of each 21-day cycle for CD30 Negative/Unknown cohort.
- CD30 Positive: Brentuximab Vedotin 1.8 mg/ kg (1.2 mg/kg in patients with grade 2 peripheral neuropathy at enrollment) administered by IV infusion given over approximately 30 minutes on Day 1 of each 21-day cycle for CD30 Positive cohort.
Period: Overall Study
Arm/Group | CD30 Negative/Unknown | CD30 Positive
Started | 11 | 7
Completed | 0 | 0
Not Completed | 11 | 7
Not completed — Death | 1 | 1
Not completed — Disease Progression | 10 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CD30 Negative/Unknown | CD30 Positive | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 7 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (9.09) | 32.2 (9.18) | 35.9 (9.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 10 | 7 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 10 | 6 | 16
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 6 | 13
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response (Percent of Patients With Complete Response or Partial Response)
Description: Measured by RECIST v1.1 and tumor markers (AFP and BhCG). CR - disappearance of all target lesions and normalization of serum tumor markers for at least 4 weeks. When only evidence of disease is elevated serum tumor markers, then values must fall below the upper limit of normal for the assay and remain at that level for at least 4 weeks. PR - at least a 30% decrease in the sum of the diameters of target lesions compared to the baseline sum diameters for at least 2 measurements 1 month apart with the serum markers as stable/decreasing. When only evidence of disease is elevated serum tumor markers, then values must fall >=90% below baseline pretreatment levels for BhCG or 50% decrease below baseline pretreatment levels for AFP and persist for 6 weeks. If both tumor markers are elevated and one falls below 90% the other should fall at least below 50% of baseline pretreatment levels.The percent of patients with objective response and its 95% exact confidence interval will be provided.
Time Frame: Up to 1 year
Population: All patients who received at least one dose of study medication and at least one evaluable assessment after treatment.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | CD30 Negative/Unknown | CD30 Positive
Number analyzed (Participants) | 10 | 6
percentage of patients | 0 [NA to NA] — There were no patients who achieved CR or PR. The confidence interval could not be estimated. | 0 [NA to NA] — There were no patients who achieved CR or PR. The confidence interval could not be estimated.

2. Secondary Outcome: Progression Free Survival
Description: Duration of time from the start of treatment to time of documented progression or death. Patients who did not progress or die were censored on their last evaluation date. Kaplan-Meier methods will be used and the median and 95% confidence intervals will be calculated.
Time Frame: Up to 2 years
Population: All patients who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CD30 Negative/Unknown | CD30 Positive
Number analyzed (Participants) | 11 | 7
months | 1.38 [0.00 to 2.07] | 1.15 [0.92 to 2.11]

3. Secondary Outcome: Overall Survival
Description: Duration of time from the start of treatment to time of death due to any causes. Patients who did not die were censored on their last known alive date. Kaplan-Meier methods will be used and the median and 95% confidence intervals will be calculated.
Time Frame: Up to 2 years
Population: All patients who received at least one dose of study medication.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | CD30 Negative/Unknown | CD30 Positive
Number analyzed (Participants) | 11 | 7
months | 5.89 [1.64 to 8.19] | 2.53 [1.12 to 12.89]

4. Secondary Outcome: Number of Patients With Treatment Related Adverse Events Grade 3 or Above
Description: Number of unique patients who had a treatment related (possible, probable or definite) adverse event with grade >= 3 using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Time Frame: Up to 2 years
Population: All patients who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | CD30 Negative/Unknown | CD30 Positive
Number analyzed (Participants) | 11 | 7
Participants | 0 | 2

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | CD30 Negative/Unknown | CD30 Positive
All-Cause Mortality (participants affected / at risk) | 8/11 | 6/7
Serious Adverse Events (participants affected / at risk) | 2/11 | 3/7
Other Adverse Events (participants affected / at risk) | 11/11 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CD30 Negative/Unknown (N=11) | CD30 Positive (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Death NOS (General disorders) | 0 | 1
Infusion related reaction (General disorders) | 0 | 1
Sudden death NOS (General disorders) | 0 | 1
Lung infection (Infections and infestations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Presyncope (Nervous system disorders) | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CD30 Negative/Unknown (N=11) | CD30 Positive (N=7)
Anemia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Hearing impaired (Ear and labyrinth disorders) | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 4 | 5
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 5 | 3
Vomiting (Gastrointestinal disorders) | 3 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 6 | 4
Infusion related reaction (General disorders) | 0 | 1
Pain (General disorders) | 3 | 1
Papulopustular rash (Infections and infestations) | 0 | 1
Cholesterol high (Investigations) | 1 | 0
Weight loss (Investigations) | 2 | 0
Anorexia (Metabolism and nutrition disorders) | 4 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Dysphasia (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 3 | 0
Nervous system disorders - Other (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 8 | 3
Anxiety (Psychiatric disorders) | 2 | 1
Depression (Psychiatric disorders) | 1 | 0
Psychiatric disorders - Other (Psychiatric disorders) | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 2
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/19/NCT02689219/Prot_SAP_000.pdf